CLINICAL TRIAL: NCT04050189
Title: Validation of the In-utero Transmission of Probiotics From the Mother to the Baby: A Randomized Crossover Pilot Study
Brief Title: Validation of the In-utero Transmission of Probiotics
Acronym: PROBIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-3242
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: In Utero Drug Exposure
Keywords: probiotic; in-utero transmission; pilot study

STUDY DESIGN:
Intervention Model Description: 2-arms randomized crossover pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prenatal probiotic (Active Comparator): will take probiotics every day from the 34th week of pregnancy until delivery; taking placebo for 10 days after delivery
  Interventions: Biological: Natural products: Probiotics; Other: Placebo
- postnatal probiotic (Active Comparator): will take placebo every day from the 34th week of pregnancy until delivery; taking probiotics for 10 days after delivery
  Interventions: Biological: Natural products: Probiotics; Other: Placebo

INTERVENTIONS:
Biological: Natural products: Probiotics — Probiotics intake every day (1.5 gram) from 34 weeks of gestation to delivery OR from delivery to 10 days postpartum
Other: Placebo — Placebo intake every day (1.5 gram) from 34 weeks of gestation to delivery OR from delivery to 10 days postpartum

SUMMARY:
This pilot project aims at confirming the in-utero transmission of probiotics, from the mother to the baby. Women aged 18 to 42 years, with a single pregnancy, considered low risk will be approached for this study. Women will take the investigational products between 34 weeks of pregnancy up to 10 days post-partum. Investigational products are probiotics (5 bacterial strains) compared to placebo.

DETAILED DESCRIPTION:
Rational: Studies have shown that probiotics given to babies can reduce perinatal complications. A change of practice should therefore be introduced in the management of premature newborns. However, one could assume that probiotic administration before birth could be as effective if not more. Indeed, one could hypothesise that when the newborn is exposed to probiotics earlier, the protective effect is potentially increased.

Objective: This pilot project aims at confirming the in-utero transmission of probiotics, from the mother to the baby.

Population: Women aged 18 to 42 years, with a single pregnancy, considered low risk will be approached for this study Products under study: Probiotics containing 5 bacterial strains (total of 12 million colony-forming unit / day) vs. Placebo.

Procedure: At 32-33 weeks, participants will complete questionnaires (medical, obstetrical, socio-demographic data) and will be randomized (double-blind) in one of the 2 following groups:

Group A: taking probiotics every day from the 34th week of pregnancy until delivery; taking placebo for 10 days after delivery.

Group B: taking placebo every day from the 34th week of pregnancy until delivery; taking probiotics for 10 days after delivery.

Follow-up: All women will complete a logbook to monitor the study products intake and monitor side effects until the end of the study (10 days postpartum).

Samples: maternal stool samples, vaginal secretions, stool (and meconium) as well as breast milk (and colostrum) will be taken at different times of the study to confirm the presence of probiotics and transmission between the mother and the baby.

ELIGIBILITY:
Inclusion Criteria:

* Women with a single pregnancy
* Women with a low risk pregnancy
* Women wishing to breastfeed at birth
* Women randomized between 32 0/7 - 33 6/7 weeks of gestation

Exclusion Criteria:

* History of obstetric complications (prematurity <37 weeks, preeclampsia , gestational diabetes treated with insulin)
* Obstetric or fetal complications known for current pregnancy such as threaten preterm labor (premature rupture of membranes or preterm labor), chorioamnionitis, placenta previa, active vaginal bleeding, cervical cerclage, fetal distress or anomalies, corticosteroid therapy
* Risk factors for obstetric complications during current pregnancy such as gestational diabetes, type I / II diabetes and high blood pressure (systole ≥140 and diastole ≥90)
* Antibiotic use within 2 weeks before randomisation
* Intake of probiotics or foods enriched with active cultures (fermented milk, kefir, kombucha ...) within 2 weeks before randomisation
* Women positive for Group B Streptococcus during previous pregnancies
* Weakened immune system (AIDS, lymphoma, chemoradiotherapy or corticotherapy, immunosuppressive pathology)
* Allergy or intolerance to lactose, soy or yeast.
* Women under Coumadin
* Women who plan to give birth outside the participating center
* Women who do not plan to breastfeed or extract their milk in the first 10 days after delivery.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
in-utero transmission of probiotic | at birth
  presence (yes or no) of probiotic (specific bacterial strains) in neonate meconium

SECONDARY OUTCOMES:
transmission of probiotic to colostrum | at birth
  presence(yes or no) of probiotic (specific bacterial strains) in colostrum
transmission of probiotic to maternal milk | 10 days postpartum
  presence (yes or no) of probiotic (specific bacterial strains) in breastmilk
transmission of probiotic to maternal vaginal tract | 37 weeks of gestation
  presence (yes or no) of probiotic (specific bacterial strains) in maternal vaginal swab
transmission of probiotic to maternal gut | 37 weeks of gestation
  presence (yes or no) of probiotic (specific bacterial strains) in maternal stools
postnatal transmission of probiotic to the neonate | 10 days postpartum
  presence (yes or no) of probiotic (specific bacterial strains) in neonate stools

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, Principal Investigator — CIUSSS-Estrie-CHUS hospital
Locations (1):
- CIUSSS de L'Estrie-CHUS Hospital, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
This is a pilot study. Samples and data will be used to confirm the principal hypothesis and explorative secondary objectives.